CLINICAL TRIAL: NCT06300398
Title: A Randomized, Double-blind, Placebo-controlled, Single and Multiple Ascending Dose Study to Investigate the Safety, Tolerability, Pharmacokinetics, Pharmacodynamics and Food Effect of IAMA-6 Administered Orally to Healthy Adults
Brief Title: IAMA-6 Oral Dose Study in Healthy Adults
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Iama Therapeutics S.r.l. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Other
Other Study IDs: ECS_IAMA23_0101
Record Dates: First submitted 2024-02-23; First posted 2024-03-08 (Actual); Last update posted 2024-03-12 (Actual); Status verified 2024-03

CONDITIONS: Neurodevelopmental Disorders
MeSH Terms: conditions — Neurodevelopmental Disorders

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Part A: Single Ascending Dose (SAD) (Experimental): Single oral doses (6 dose cohorts) of IAMA-6 liquid suspension or placebo-to-match IAMA-6 liquid suspension in fasted participants
  Interventions: Drug: IAMA-6; Drug: Placebo
- Part B: Food Effect (FE) (Experimental): Single oral dose (1 dose cohort) of IAMA-6 liquid suspension in fed participants
  Interventions: Drug: IAMA-6
- Part C: Multiple Ascending Dose (MAD) (Experimental): Multiple oral doses (3 dose cohorts) of IAMA-6 liquid suspension or placebo-to-match IAMA-6 liquid suspension for 7 days in fasted or fed participants
  Interventions: Drug: IAMA-6; Drug: Placebo

INTERVENTIONS:
Drug: IAMA-6 — IAMA-6 liquid suspension
Drug: Placebo — Placebo-to-match IAMA-6 liquid suspension
  Arms: Part A: Single Ascending Dose (SAD); Part C: Multiple Ascending Dose (MAD)

SUMMARY:
The main purpose of this study is to evaluate the safety, tolerability, pharmacokinetics, pharmacodynamics and food effect of IAMA-6 administered orally to healthy adults.

DETAILED DESCRIPTION:
The Sponsor's proposed clinical trial is a randomized, double blind, placebo controlled first in human study. This is a single ascending dose (SAD) and multiple ascending dose (MAD) study to investigate the safety, tolerability, pharmacokinetics, pharmacodynamics and food effect of IAMA-6 administered orally to healthy adults.

The study consists of the following 3 elements:

Part A: Single Ascending Dose

Part A includes up to 6 cohorts of 8 healthy male and female participants, each receiving a single oral dose of IAMA-6 or placebo (6 IAMA-6 and 2 placebo):

1. Group A1 (N=8): IAMA-6 Dose 1 (N=6) or Placebo (N=2)
2. Group A2 (N=8): IAMA-6 Dose 2 (N=6) or Placebo (N=2)
3. Group A3 (N=8): IAMA-6 Dose 3 (N=6) or Placebo (N=2)
4. Group A4 (N=8): IAMA-6 Dose 4 (N=6) or Placebo (N=2)
5. Group A5 (N=8): IAMA-6 Dose 5 (N=6) or Placebo (N=2)
6. Group A6 (N=8): IAMA-6 Dose 6 (N=6) or Placebo (N=2)

In each cohort, treatment will be randomly assigned, such that 2 participants (1 IAMA-6 and 1 placebo) will be dosed first, as sentinel subjects. If safety and tolerability results are acceptable, based on any adverse reactions or events, after at least 24 hours, the remaining 6 participants will be randomly assigned treatment (5 IAMA-6 and 1 placebo) and dosed. All doses will be taken in a fasting state.

Dose escalation will only occur after all safety data from the completed dose group have been reviewed by the sponsor and site investigator, and it has been determined safe to proceed to the next dose cohort.

Part B: Food Effect After completion of the SAD dose escalation (Part A and review of the PK and safety data, one cohort of subjects who received IAMA-6 (n = 6) at the highest safe dose with measurable exposure, will return to the clinic to receive a 2nd dose of IAMA-6 in the fed state to determine the potential effect of food on the bioavailability of IAMA-6 before initiating Part C. The dose of IAMA-6 will be taken after a high fat meal as described in regulatory guidelines (FDA model).

Part C: Multiple Ascending Dose Part C includes up to 3 cohorts of 8 healthy male and female participants, each receiving oral doses of IAMA-6 or placebo (6 IAMA-6 and 2 placebo) for 7 consecutive days, as follows, the doses and the posology being selected according to their acceptable safety, tolerability and pharmacokinetics in Part A. Doses will be taken either with or without food according to the results of Part B of the study.

1. Group C1 (N=8): IAMA-6 Dose X (N=6) or Placebo (N=2)
2. Group C2 (N=8): IAMA-6 Dose Y (N=6) or Placebo (N=2)
3. Group C3 (N=8): IAMA-6 Dose Z (N=6) or Placebo (N=2)

In each cohort, treatment will be randomly assigned, such that 2 participants (1 IAMA-6 and 1 placebo) will be dosed first, as sentinel subjects. If the safety and tolerability results are acceptable, based on any reaction or adverse events, after at least 72 hours, the 6 remaining participants will be randomly assigned treatment (5 IAMA-6 and 1 placebo) and dosed. There will be a 7 day follow up after last dosing for all participants followed by review of clinical and laboratory safety data before starting treatment of the next dose cohort.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male and female subjects.
* Aged between 18 and 55 years.
* Written informed consent; willing and able to comply with procedures.
* Females will not be pregnant or lactating, and females of childbearing potential and males will agree to use contraception.
* Body mass index of 18.0 to 30.0 kg/m2, inclusive; and a total body weight >50 kg up to a maximum of 110 kg.
* The subject must be willing to return to the study centre for study treatment and study-related follow-up procedures as required by the protocol.

Exclusion Criteria:

* Current or past history of a clinically significant (as judged by the Investigator) cardiovascular, cerebrovascular, respiratory, gastrointestinal, hematologic, renal, hepatic, immunologic, metabolic, urologic, neurologic, dermatologic, psychiatric, or other major disease/condition, as determined by the Principal Investigator or Designee.
* Any history of central nervous system problems (e.g. epilepsy, head injury, loss of consciousness).
* Any history of malignancy in the previous 5 years involving any organ system (other than localised basal cell carcinoma of the skin).
* Body Mass Index: <18 kg/m2 , or >30 kg/m2.
* Abnormal vital signs, including known history of hypertension, resting oxygen saturation <95% by pulse oximetry.
* ECG at screening or on Day -1 showing QTcF interval >450 msec in males or >470 msec in females, or presence of any clinically significant dysrhythmia.
* History of hypersensitivity to any medicinal product(s) or severe hypersensitivity/anaphylaxis with unclear aetiology.
* Any clinically significant abnormal chemistry values.
* Any clinically significant abnormal haematology values.
* Blood donation within the past 3 months.
* Seropositivity for HBsAg, HCV, HIV 1, or HIV 2.
* Has a positive nasopharyngeal test for SARS-CoV-2 within 48h before unit admission.
* If female, has a positive highly sensitive urine pregnancy test at Screening or Day 1.
* If female and of child-bearing potential, and not meeting the approved criteria for highly effective methods of birth control.
* Receipt of any Investigational Drug within the past 6 months.
* Use of prescription medication within 14 days prior to dosing and antibiotics within 30 days prior to dosing.
* Intake of OTC preparations, vitamins, minerals, herbal remedies within 48h prior to dosing.
* Current smokers or history of smoking in previous 6 months.
* Current or history of drug, alcohol, nicotine abuse, or excessive coffee (>5 cups/day) or tea drinking (>5 cups/day).
* Inadequate comprehension of study risks and requirements.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 72 (Estimated)
Dates: Start 2024-01-08 (Actual); Primary Completion 2024-09 (Estimated); Study Completion 2024-09 (Estimated)

PRIMARY OUTCOMES:
Number of participants with adverse events (AEs) | From time of the first dose to study completion, an average of 1 year
  All AEs will be coded by Medical Dictionary for Regulatory Activities (MedDRA; Version 26.1 or later) System Organ Class and Preferred Term. The incidence of the following events will be summarized by treatment group and study part (i.e. Part A, Part B and Part C):
  * Treatment-emergent AEs (TEAEs).
  * TEAEs by severity.
  * TEAEs by causality.
  * Serious TEAEs.
Number of participants with serious adverse events (SAEs) | From time of the first dose to study completion, an average of 1 year
  All AEs will be coded by Medical Dictionary for Regulatory Activities (MedDRA; Version 26.1 or later) System Organ Class and Preferred Term. The incidence of the following events will be summarized by treatment group and study part (i.e. Part A, Part B and Part C):
  * Treatment-emergent AEs (TEAEs).
  * TEAEs by severity.
  * TEAEs by causality.
  * Serious TEAEs.
Number of participants with physical examination abnormalities | Part A: Baseline and Day 8; Part B: Day 8; Part C: Baseline and Day 14
  Physical examinations and mean changes from baseline (when applicable) will be descriptively summarized by treatment group and study part (i.e. Part A, Part B and Part C).
Number of participants with vital sign abnormalities | Part A: Baseline and Days 1, 2 and 8; Part B: Days 1, 2 and 8; Part C: Baseline and Days 1-8 and 14
  Vital sign parameters and mean changes from baseline (when applicable) will be descriptively summarized by treatment group and study part (i.e. Part A, Part B and Part C).
Number of participants with electrocardiogram (ECG) abnormalities | Part A: Baseline and Days 1, 2 and 8; Part B: Days 1, 2 and 8; Part C: Baseline and Days 1-8 and 14
  Electrocardiogram measurements and mean changes from baseline will be descriptively summarized by treatment group and study part (i.e. Part A, Part B and Part C).
Number of participants with clinical laboratory abnormalities | Through study completion, an average of 1 year
  Clinical laboratory test parameters and mean changes from baseline will be descriptively summarized by treatment group and study part (i.e. Part A, Part B and Part C).
Number of participants with hearing abnormalities | Part C: Screening and Day 6
  The results of the hearing tests (Part C) will be descriptively summarized by timepoint and the change vs baseline (when applicable) will also be analysed.
  Hearing tests performed: High Frequency Audiometry (HFA) and Pure Tone Audiometry (PTA).

SECONDARY OUTCOMES:
Cmax pharmacokinetic (PK) parameter of IAMA-6 following single and multiple oral doses | Parts A and B: Day 1, Day 2 and Day 3; Part C: Day 1 Day 2, Day 7, Day 8 and Day 9
  Pharmacokinetic concentrations and/or parameters will be summarized using descriptive statistics by treatment arm and study part (i.e. SAD/MAD).
Tmax pharmacokinetic (PK) parameter of IAMA-6 following single and multiple oral doses | Parts A and B: Day 1, Day 2 and Day 3; Part C: Day 1 Day 2, Day 7, Day 8 and Day 9
  Pharmacokinetic concentrations and/or parameters will be summarized using descriptive statistics by treatment arm and study part (i.e. SAD/MAD).
T1/2 pharmacokinetic (PK) parameter of IAMA-6 following single and multiple oral doses | Parts A and B: Day 1, Day 2 and Day 3; Part C: Day 1 Day 2, Day 7, Day 8 and Day 9
  Pharmacokinetic concentrations and/or parameters will be summarized using descriptive statistics by treatment arm and study part (i.e. SAD/MAD).
AUC(0-t) and AUCτ pharmacokinetic (PK) parameters of IAMA-6 following single and multiple oral doses | Parts A and B: Day 1, Day 2 and Day 3; Part C: Day 1 Day 2, Day 7, Day 8 and Day 9
  Pharmacokinetic concentrations and/or parameters will be summarized using descriptive statistics by treatment arm and study part (i.e. SAD/MAD).
Vd pharmacokinetic (PK) parameters of IAMA-6 following single and multiple oral doses | Parts A and B: Day 1, Day 2 and Day 3; Part C: Day 1 Day 2, Day 7, Day 8 and Day 9
  Pharmacokinetic concentrations and/or parameters will be summarized using descriptive statistics by treatment arm and study part (i.e. SAD/MAD).
CL pharmacokinetic (PK) parameters of IAMA-6 following single and multiple oral doses | Parts A and B: Day 1, Day 2 and Day 3; Part C: Day 1 Day 2, Day 7, Day 8 and Day 9
  Pharmacokinetic concentrations and/or parameters will be summarized using descriptive statistics by treatment arm and study part (i.e. SAD/MAD).
λz pharmacokinetic (PK) parameters of IAMA-6 following single and multiple oral doses | Parts A and B: Day 1, Day 2 and Day 3; Part C: Day 1 Day 2, Day 7, Day 8 and Day 9
  Pharmacokinetic concentrations and/or parameters will be summarized using descriptive statistics by treatment arm and study part (i.e. SAD/MAD).
Urine volume | Before treatment (Day -1) and after treatment (Day 1 in Part A and Day 7 in Part C) for a 24-hour period
  Urine volume will be summarized using descriptive statistics by treatment arm and study part (i.e. SAD/MAD).
Na+ excretion | Before treatment (Day -1) and after treatment (Day 1 in Part A and Day 7 in Part C) for a 24-hour period
  Urinary sodium concentration will be summarized using descriptive statistics by treatment arm and study.
K+ excretion | Before treatment (Day -1) and after treatment (Day 1 in Part A and Day 7 in Part C) for a 24-hour period
  Urinary potassium concentration will be summarized using descriptive statistics by treatment arm and study.
Sleep assessment | Day 2 (Parts A, B, C), Days 8 and 9 (Part C)
  Sleep assessment using the Leeds Sleep Evaluation Questionnaire (LSEQ). Score between 0 and 100 for each question (total of 10 questions). Higher scores mean a worse outcome.
  The results of the questionnaire will be descriptively summarized by timepoint and the change vs baseline (when applicable) will also be analysed.

CONTACTS AND LOCATIONS:
Overall Officials: Stefano Milleri, MD, Principal Investigator — Centro Ricerche Cliniche di Verona srl
Locations (1):
- Centro Ricerche Cliniche Di Verona S.r.l., Verona, Italy

IPD SHARING:
Plan to Share IPD: No